CLINICAL TRIAL: NCT00054054
Title: Docetaxel (NSC-628503), Cisplatin (NSC-119875), And 5-Fluorouracil (NSC-19893) Induction Chemotherapy Followed By Accelerated Fractionation/Concomitant Boost Radiation And Concurrent Single Agent Cisplatin (NSC-119875), In Patients With Advanced Squamous Cell Head And Neck Cancer
Brief Title: S0216, Combination Chemotherapy and RT in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Laurence H. Baker, D.O., Southwest Oncology Group-Group Chair's Office
Purpose: Treatment
Other Study IDs: CDR0000269781; S0216 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival of patients with stage III or IV squamous cell head and neck cancer treated with docetaxel, cisplatin, and fluorouracil followed by accelerated fractionation/concomitant boost radiotherapy and cisplatin.
* Determine the unconfirmed complete response rate in these patients after treatment with induction chemotherapy.
* Determine the overall complete response rate (confirmed and unconfirmed) in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE:

* Induction Chemotherapy: Patients receive docetaxel IV over 1 hour and cisplatin IV over 30-60 minutes on day 1 and fluorouracil IV continuously on days 1-4. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity.
* Chemoradiotherapy: Beginning within 3-4 weeks after administration of the second course of induction chemotherapy, patients receive accelerated fractionation radiotherapy once daily, 5 days per week, for 6 weeks with concomitant boost radiotherapy once daily, 5 days a week, for the last 2.5 weeks of radiotherapy. Patients also receive concurrent cisplatin IV over 30-60 minutes on days 1 and 22.

Patients are followed every 2 months for 1 year, every 3 months for 2 years, every 4 months for 1 year, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck (excluding lip, nasopharynx, paranasal sinus, and salivary gland) by biopsy or fine needle aspirate of the primary lesion or neck mass

  * Stage III or IV disease
* No evidence of distant metastases

  * Negative chest x-ray
* Primary site in the head and neck region must be identified

  * No unknown primary site
* Considered to be appropriate for definitive radiotherapy with curative intent

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase less than 2 times ULN
* ALT or AST less than 1.5 times ULN

Renal

* Creatinine less than 1.5 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No unstable or uncontrolled angina

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* No evidence of pre-existing peripheral neuropathy
* No active systemic infection
* No history of hypersensitivity reaction to products containing polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy

Surgery

* No prior surgery for head or neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Study Chair — The Cleveland Clinic
Locations (95):
- United States (94):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center, Fresno, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Veterans Affairs Medical Center - Salisbury, Salisbury, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Adelstein DJ, Moon J, Hanna E, Giri PG, Mills GM, Wolf GT, Urba SG. Docetaxel, cisplatin, and fluorouracil induction chemotherapy followed by accelerated fractionation/concomitant boost radiation and concurrent cisplatin in patients with advanced squamous cell head and neck cancer: A Southwest Oncology Group phase II trial (S0216). Head Neck. 2010 Feb;32(2):221-8. doi: 10.1002/hed.21179. PMID 19557750
- [Result] Adelstein DJ, Moon J, Hanna E, et al.: S0216: a Southwest Oncology Group (SWOG) phase II trial of docetaxel (T), cisplatin (P), and fluorouracil (F) induction followed by accelerated fractionation/concomitant boost (AF/CB) radiotherapy (RT) and concurrent cisplatin for advanced head and neck squamous cell cancer (HNSCC). [Abstract] J Clin Oncol 25 (Suppl 18): A-6014, 302s, 2007.